CLINICAL TRIAL: NCT04215107
Title: Fetal Distribution of Feto-placental Blood Flow Related to Placental Nutrient Transport and Maternal Food Intake
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guttorm Haugen (Other)
Responsible Party: Sponsor-Investigator, Guttorm Haugen, Clinical Professor, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: REK ref: 2018/1034B
Record Dates: First submitted 2019-03-04; First posted 2020-01-02 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Fetal Growth Restriction
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Crossover study Group. Each patient will be examined 2 seperate days. Randomized to standard breakfast meal or prolonged fasting. The examinator will be blinded to patient meal status.
  Interventions: Other: Standard breakfast meal
- IUGR group (Other): Will only be examined one day. First ultrasound during fasting, and the second ultrasound 2 hours after a standard breakfast meal.
  Interventions: Other: Standard breakfast meal

INTERVENTIONS:
Other: Standard breakfast meal — The first ultrasound will be preformed during fasting. IUGR group will be served a standard breakfast meal, and perform the second ultrasound after 2 hours from the meal.
  The control group will be crossover randomized to meal or prolonged fasting. It will be performed 4 ultrasounds: during fasting and 2 hours after standard breakfast meal. During fasting and during prolonged fasting.

SUMMARY:
Aims

The primary aim is to examine the relation between maternal nutrition, placental transport of nutritional substances, and fetal blood flow distribution in normal pregnancies and in pregnancies complicated by altered fetal growth. Specific aims:

1. Examine the relation between fetal glucose, amino acid and lipid consumption, and ultrasound Doppler measures of fetal cerebral vascular resistance.
2. Examine the influence of extended fasting for two hours compared to a standard meal in a group with appropriate fetal group on fetal liver blood flow and fetal cerebral vascular resistance. The examinations will be performed at approximately 36 weeks gestation.
3. Examine the influence of a standard maternal meal on fetal liver blood flow and fetal cerebral vascular resistance in pregnancies complicated by fetal growth restriction (FGR).

Study 1: Investigator will use the 130 fetal-maternal pairs from the "placental 4 vessel sampling method" (see below) which includes measures on fetal blood flow distribution. Some calculations will be performed on the restricted cohort of 70 pregnancies who also includes maternal blood flow measures.

Study 2: A limitation of investigators previous studies on the influence of glucose intake or a regular maternal meal on fetal blood flow distribution in healthy pregnancies with appropriate fetal growth is the lack of a control group without food intake (extended fasting for two hours). To serve as participants own control the included participants will meet for examinations at two different days (one with food intake and one with extended fasting) within a few days interval. Participants will be examined in the morning and two hours after food intake or after two hours extended fasting. The study will include 25 pregnancies with gestational age about 36 weeks

Study 3: Investigator will include approximately 55 women (see power calculation below) with pregnancies complicated by FGR defined as estimated birth weight (EFW) below the 3rd percentile and/or EFW below the 10th percentile and sign of fetal Doppler blood flow redistribution representing possible fetal compromise . Investigator hypothesize that there will be no reduction in fetal cerebral vascular resistance (measured as change in MCA-PI from before to after food intake). Fetal liver blood flow will also be measured.

Methods The "Placental 4 vessel sampling method" This method has recently been developed by investigators research group and described in recent publications. In brief, blood samples are obtained from incoming (arterial) and outgoing (venous) vessels both at the maternal and fetal side of the placenta simultaneously during cesarean section. Samples have been taken from women with normal pregnancies but with a range of BMI and metabolic profiles: the physiological range group (undergoing cesarean delivery on own request).

Investigators have a complete dataset including blood sampling and fetal blood flow measurements in the UV, DV and MCA-PI in 130 women. Further, investigators have maternal blood flow measures in 70 of these pregnancies.

Doppler blood flow measurements Doppler blood flow measurements will be performed in the morning immediately before (fasting state) and after a standard breakfast meal (SBM) (approximately120 min). Internal vessel diameter (D) and time-averaged maximum velocity (TAMX) will be measured in the straight portion of the intra-abdominal UV and at the inlet of DV, respectively.

In the MCA Doppler velocity waveforms are sampled from the proximal part emerging from the circle of Willis . MCA in the hemisphere near the transducer will be used unless there are better insonation properties in the opposite hemisphere. Umbilical artery Doppler traces will be sampled in a free-floating loop. The Doppler tracings will be used to measure fetal heart rate (FHR). All measurements will be performed during periods of fetal quiescence.

ELIGIBILITY:
Inclusion Criteria:

* Control group: Pregnant caucasian women With singleton fetus, and without any disease which can influence placental function

Exclusion Criteria:

* Food allergy
* use of medicine which can influence placental function

Ages: 16 Years to 58 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-10-11 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Doppler measures of fetal cerebral vascular resistance as mean cerebral artery pulsatility index (MCA-PI) | 2-2,5 years
  Examine the influence of extended fasting for two hours compared to a standard meal in a group with appropriate fetal group on fetal cerebral vascular resistance, measured as MCA-PI, ranging from 1,2-2,5. Values below 1,1 represent poor outcome. The examinations will be performed at approximately 36 weeks gestation.
  Examine the influence of a standard maternal meal on fetal cerebral vascular resistance, measured as MCA-PI, in pregnancies complicated by fetal growth restriction (FGR).
Doppler measures of fetal liver blood flow (ml/min) | 2-2,5 years
  Examine the influence of extended fasting for two hours compared to a standard meal in a group with appropriate fetal group on fetal liver blood flow (ml/min) .The examinations will be performed at approximately 36 weeks gestation.
  Examine the influence of a standard maternal meal on fetal liver blood flow (ml/min) pregnancies complicated by fetal growth restriction (FGR).
Examine the relation between nutrient (glucose, amino acid and lipid) transfer to the fetus (mmol/ml), and ultrasound Doppler measures of fetal cerebral vascular resistance, measured as MCA-PI (mean cerebral artery pulsatility index | 1 year
  Investigators will use the 130 fetal-maternal pairs from the "placental 4 vessel sampling method". In brief, blood samples are obtained from incoming (arterial) and outgoing (venous) vessels both at the maternal and fetal side of the placenta simultaneously during cesarean section. Nutrient concentration is measured as mmol/ml. This sample also includes doppler measures of blood flow (ml/min) in the umbilical vein (fetal side) and in the uterine artery (maternal side), and mean cerebral artery pulsatility-index (MCA-PI) which is a measurement for cerebral vascular resistance.
  The absolute transfer of the nutrients to the fetus is measured in mmol/min, by combining blood flow (ml/min) and nutrient concentration (mmol/ml). Investigator will examine the correlation between absolute fetal nutrients transfer (mmol/ml) and fetal cerebral vascular resistance (MCA-PI).

CONTACTS AND LOCATIONS:
Overall Officials: Guttorm Haugen, Principal Investigator
Locations (1):
- Oslo university hospital, Oslo, Norway